CLINICAL TRIAL: NCT06443840
Title: AUTONHOME: Impact of a Self-rehabilitation and Tele-rehabilitation Program on the Post-stroke Care Pathway : Preliminary Study
Brief Title: Impact of a Self-rehabilitation and Tele-rehabilitation Program on the Post-stroke Care Pathway
Acronym: AUTONHOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association APPROCHE (Other)
Collaborators: Société Neuradom (Unknown); IMT Atlantique Brest (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-A01298-37
Record Dates: First submitted 2024-05-14; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Hemorrhagic Unilateral Cortico-subcortical Hemispheric Stroke; Ischemic Stroke
Keywords: post-stroke; tele-rehabilitation; self-rehabilitation; AutonHome; medical device; Physical Medicine and Rehabilitation; Rehabilitation Medicine
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This protocol is carried out in accordance with the European Regulation 2017/745 on Medical Devices (MDR) and concerns a Class I medical device (MD) of category 4.2 (Article 82 MDR), corresponding to the CE marked MD used for its intended purpose without the objective of establishing conformity, and with an additional non-invasive and non-burdensome procedure.
  This is a comparative, prospective, multicenter study (4 centers), controlled, randomized, open-label, with 2 parallel arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants will be randomised into a control group, undergoing conventional in-centre rehabilitation.
- Experimental group (Experimental): The experimental group will have to carry out the programme of self-rehabilitation and tele-rehabilitation with the AutonHome® device in addition to conventional rehabilitation.
  Interventions: Device: AutonHome® device

INTERVENTIONS:
Device: AutonHome® device — The experimental group will have to carry out the programme of self-rehabilitation and tele-rehabilitation with the AutonHome® device in addition to conventional rehabilitation.
  Arms: Experimental group

SUMMARY:
The AutonHome® clinical investigation, proposed by Dr Charles FATTAL (coordinator of this study), and carried out by the Association Approche (delegated promoter), aims to use the AutonHome® selfeducation device for the rehabilitation of patients who have suffered a Cerebrovascular Accident (CVA), and thus respond to the problems of therapeutic discontinuity highlighted today. Neuradom's AutonHome® device combines self-education and telecare. This device makes it possible to carry out personalised self-education programmes supervised by the therapist, enabling the therapeutic link with the patient to be maintained without the need for the patient to travel. This tool has already proved its usability and perceived usefulness in a previous clinical study, which demonstrated the feasibility of a self-education programme for hemiplegic patients, based on feedback. AutonHome® was considered by users to be a relevant, useful and safe complement to conventional rehabilitation.

On the basis of this feasibility study, the investigators wished to develop a second study around this AutonHome® device. In this second clinical investigation, in addition to perceived usefulness, the main objective is to demonstrate, in a population of stroke victims, that an experimental care pathway combining supervised self-education via AutonHome® with conventional re-education optimises the care pathway in terms of sensory-motor recovery, but also in terms of reduced length of stay and functional and medico-economic added value.

This clinical trial involves two parallel arms. Participants will be randomised into a control group, undergoing conventional in-centre rehabilitation, or into an experimental group, with self-rehabilitation and tele-rehabilitation in addition to conventional rehabilitation. The AutonHome study is a pilot study, with the aim of including 40 participants. Each centre will recruit 10 participants on a 1:1 randomisation basis, with 5 in the experimental group and 5 in the control group. Participants will be monitored for 15 weeks. This clinical investigation is multicentre, with 4 centres involved: the Centre Bouffard Vercelli (66962, Perpignan), the CMRRF de Kerpape (56275 Ploemeur), the association Saint-Hélier (35043, Rennes), and the Fondation ILDYS (29684 Roscoff).

ELIGIBILITY:
Inclusion Criteria:

* Participants who signed the written consent form to participate in the study after free and informed information
* Participants affiliated to a social security scheme (beneficiary or beneficiary) outside the AME.
* 18 years ≤ age ≤ 85 years,
* 1st recent ischemic or hemorrhagic unilateral cortico-subcortical hemispheric stroke
* Minimum post-stroke delay: 7 days
* Maximum post-stroke delay : 30 days
* SOFMER category 2: moderate strokes called category 2 according to SOFMER with an NIHSS (initial score of the National Institute of Health Stroke Scale) between 5 and 14 (Several deficiencies or motor deficit of the lower limb prohibiting walking, with recovery potential, a probable autonomy project (unilateral stroke).
* MoCA > 23

Exclusion Criteria:

* Participant deprived of liberty (by judicial or administrative decision)
* Adult participant subject to a legal protection measure or unable to express their consent
* Participation in another ongoing clinical trial
* Pregnant or breastfeeding women or women of childbearing age without effective contraception
* Lack of command of the oral and written French language
* Pre-existing neurological pathology
* Severe expression disorders (expression aphasia) affecting intelligibility
* Severe comprehension disorders (comprehension aphasia)
* Major cognitive disorders of the dementia or post-dementia type
* Unstable psychiatric disorders
* Unstabilized medical pathology
* Unbalanced epilepsy
* Color blindness

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the non-inferiority of the experimental course of care, on the technical platform and at home, on the evolution of sensory-motor recovery, compared to the control course. | At 0 and 6 weeks
  Change in Fugl-Meyer score between inclusion on Day 0 and the visit on Day 45 (Week 6) Minimum = 0 Maximum = 100
  However, as an exploratory secondary endpoint (objective 1a), the sub-scores for the upper limb (UL) and lower limb (LL) will be studied separately, as well as changes at 12 weeks (D80) and 15 weeks (D105).
  * Upper limb / 66
  * Lower limb / 34 Total / 100
  The higher the Fugl Meyer score, the better the sensory-motor recovery. The Fugl Meyer scores will then be compared between the experimental course (on the technical platform and at home) and the control course.

SECONDARY OUTCOMES:
Evaluate the recovery of overall functional independence. | At 0, 6, 12 and 15 weeks
  Functional independence measure - MIF
  Independence :
  7: Complete independence (appropriate to circumstances and safe) 6: Modified independence (device, adaptation)
  Modified dependence :
  5: Supervision 4: Minimal assistance (autonomy = 75% +) 3 : Average assistance (autonomy = 50% +)
  Complete dependence 2 : Maximum assistance (autonomy = 25% +)
  If an item cannot be checked, tick level 1.
  At the end of the test, we obtain a score ranging from 18 to 126. The lower the score, the greater the disability.
The recovery of a seated and standing postural balance, walking and mobility on the plane. | At 0, 6, 12 and 15 weeks
  Berg balance scale :
  The Berg balance assessment scale was developed to measure static and dynamic balance in adults.
  This scale comprises 14 tasks rated from 0 to 4, assessing both static and dynamic balance. The total score ranges from 0 to 56 points. The higher the score, the better the assessment of balance.
The recovery of a seated and standing postural balance, walking and mobility on the plane. | At 0, 6, 12 and 15 weeks
  6min walk test (6MWT) : The six-minute walk test (6MWT) is an objective assessment of functional physical ability. It measures the distance covered by the patient when walking briskly for 6 minutes.
  The 6MWT provides a global assessment of various organ functions, in particular the cardiopulmonary, vascular and neuromuscular systems.
  Distance covered: The distance covered during the test is the main parameter measured. In general, a longer distance indicates better functional capacity. Here are some approximate reference values:
  Normal: Approximately 400 to 700 metres. Poor: Less than 300 metres. Very good: Over 800 metres.
The recovery of a seated and standing postural balance, walking and mobility on the plane. | At 0, 6, 12 and 15 weeks
  10-metre walk test (10MWT) : The 10-metre walk test is an assessment tool that measures a patient's walking speed.
  It aims to calculate the speed at which a patient can walk a distance of 10 metres.
  The walking speed obtained can be used to classify the patient into different categories:
  Less than 0.4 m/s: Walking at home. Between 0.4 and 0.8 m/s: Limited walking in the community. More than 0.8 m/s: Unlimited walking in the community.
Achievement of objectives | At 0, 6, 12 and 15 weeks
  GAS (Goal Attainment Scaling) :
  The GAS is a tool for defining specific, individualised objectives for each patient. These objectives are then evaluated in a standardised way, allowing statistical analysis of the results.
  At least 3 objectives are set and scored between -3 (regression), -2 (much less), -1 (a little less), 0 (expected result), +1 (a little more), +2 (much more).
Autonomy and social participation | At 0, 6, 12 and 15 weeks
  IPA Scale (Impact on Participation and Autonomy Questionnaire) :
  * Level of participation perceived by the participant through 32 items spread over 5 domains related to autonomy in activities inside the home (7 items), family roles (7 items), activities outside (5 items), social life and relationships (7 items), work and education (6 items). The last 6 are excluded. Score from 0 (very low level of participation) to 4 (very high level).
  * Level of perception of participation restriction: Score of 0 (major problem), 1 (minor problem), 2 (no problem).
The risk of adverse effects | Every day during 15 weeks
  Number of falls
The risk of adverse effects | Every day during 15 weeks
  Number of moderate or serious adverse events during the session
The risk of adverse effects | Every day during 15 weeks
  Visual Analog Pain Scale: Intensity and sites of pain before or during and after the session
The perception of the effort at each session | Every day during 15 weeks
  Borg scale :
  The Borg scale is generally rated from 6 to 20. The higher the number, the more intense the perceived effort.
The perceived experience of the session. | Every day during 15 weeks
  Perceived experience of the rehabilitation session in response to the following 4 questions with a scoring that comes in 5 different levels depending on the question :
  What is the patient's perception of the rehabilitation session offered? Very poor - Poor - No effect - Positive - Very positive
  What is the patient's perception of the quality of the exercises proposed? Very poor - Poor - No effect - Positive - Very positive
  What is the patient's perception of the intensity of the exercises proposed? Very poor - Poor - No effect - Positive - Very positive
  What is the patient's perception of the motivating nature of the exercises proposed? Very poor - Poor - No effect - Positive - Very positive
The perceived experience of the session. | Every day during 15 weeks
  SIMS MOTIVATION Scale ("Situation Motivation Scale") :
  The aim is to determine which type of motivation regulates an individual's behaviour during an activity.
  16 items are evaluated: Items 1, 5, 9 and 13 relate to intrinsic motivation (best type of regulation, strong feeling of autonomy).
  Items 2, 6, 10 and 14 relate to identified regulation (good type of regulation, high sense of autonomy).
  Items 3, 7, 11 and 15 refer to external regulation (poor type of regulation, low sense of autonomy).
  Items 4, 8, 12 and 16 relate to motivation (no regulation).
Compliance with and duration of sessions and stays. | Every day during 15 weeks
  Compliance (present at the session) : Yes/No
Compliance with and duration of sessions and stays. | Every day during 15 weeks
  Duration of each session (in minutes)
Compliance with and duration of sessions and stays. | Every day during 15 weeks
  Duration of stay in complete hospitalisation (in days)
Compliance with and duration of sessions and stays. | Every day during 15 weeks
  Duration of stay in partiel hospitalisation (in days)
Compliance with and duration of sessions and stays. | Every day during 15 weeks
  Duration of use at home (in days)
Study the medium-term appropriation of the selfrehabilitation system by the participants. | At 0, 6, 12 and 15 weeks
  SUS (System Usability Scale) : only for the experimental groups. The SUS consists of 10 questions in the form of statements. Each question uses a Likert scale, where the user chooses between 5 possible answers, ranging from 'Strongly disagree' to 'Strongly agree'. The answers to the 10 questions are used to construct a satisfaction score, ranging from 1 to 100. In general, a score of 75 or more is considered 'good', while between 50 and 75 it is considered 'fair' or 'correct'. A score of less than 50 indicates major problems in terms of customer satisfaction.
Compare the costs of the experimental care pathway to the costs of a conventional care pathway | Every day during 15 weeks
  Study of direct and indirect costs

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Fondation Ildys, Brest, Brittany Region
  - CMRRF de Kerpape, Ploemeur, Brittany Region
  - Association Saint-Hélier, Rennes, Brittany Region
  - Centre Bouffard Vercelli - USSAP, Perpignan, Pyrénées-Orientales

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] RAOULT, Bérengère, PONTIER, Joanna, FICHEUX, Gilles and FATTAL, Charles, 2020. Étude de faisabilité d'un parcours d'auto-rééducation de patients hémiplégiques. Kinésithérapie Scientifique. Décembre 2020. No. 626, p. 5-13.